CLINICAL TRIAL: NCT06404216
Title: The Effect of a Nordic Walking Group Training on the Physical and Mental Health of Older Adults Evacuated From Their Homes to Haifa- A Pilot Study
Brief Title: Nordic Walking Training Program for Sustaining Independent Walking in Older Adult Evacuees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Hilla Sarig Bahat, Dr., University of Haifa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSBahat
Record Dates: First submitted 2024-04-22; First posted 2024-05-08 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2024-06

CONDITIONS: Aging; Mental Health Issue; War-Related Trauma
MeSH Terms: conditions — War-Related Injuries

STUDY DESIGN:
Intervention Model Description: One arm of treatment in a special displaced population during war. This is a pilot feasibility study, prior to a full RCT in order to evaluate this protocol.
  Intervention of 2 weekly sessions for 8 weeks (total 16). Assessments will be conducted by a blinded assessor at baseline, end of training, 2+4 months post-intervention.
Masking Description: The assessor will be external, not part of the training team, to avoid bias due to trainer/therapist- training participant subjective biases.
  Therefore there is assessor blinding but not to allocation as there is one arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nordic walking group training (Experimental): The intervention will consist of 60-minute NW group sessions, twice weekly, for two months (total 16 sessions). Participants will be provided with NW sticks to use during the sessions. Each session will be led by a qualified healthcare professional that received 4 hours NW guidance qualification, and participated in 4 sessions prior to leading one. Current qualified healthcare professionals are 2 physiotherapists, and a certified nurse. Final year physiotherapy students will assist, hence each session will be guided by two members of the research team- a clinician and a student.
  A social worker will participate in one weekly session aiming to empower the participants and utilize group dynamics techniques to promote successful continuation of independent walking following the guided period.
  Interventions: Other: Nordic walking group training

INTERVENTIONS:
Other: Nordic walking group training — 16 60-minute NW group sessions, twice weekly. Sessions will be led by a qualified healthcare professional and a graduating student.
  A social worker (SP) will participate in one weekly session aiming to empower the participants and utilize group dynamics techniques to promote successful continuation of independent walking following the guided period.
  Communication throughout the study will be conducted via a WhatsApp forum, to motivate and sustain regular walking during and after the training period. Following 2 months of guidance the group will be launched independently, while keeping remote contact. Same frequency and schedule will be encouraged.

SUMMARY:
Abstract:

The purpose of this pilot study is to examine the effect and feasibility of a Nordic walking group training intervention on the physical and mental health of older adults evacuated from their homes to Haifa.

Participants:

The study will include 31 participants aged 65 and over who are in stable health and have been cleared by their physician to participate in this NW program.

Intervention:

The intervention will consist of two 60-minute Nordic walking (NW) sessions per week for two months, 16 sessions in total. Participants will be provided with walking sticks to use during the sessions. The sessions will be led by certified health professionals (PT, RN), assisted by trained undergraduate and graduate physiotherapy students.

Outcomes:

The primary outcome will be endurance to the walking sessions, and average weekly and monthly number of steps, measured by a smartphone application. Secondary outcomes will include three physical tests: 30-second sit-to-stand test, 4-meter walk test and heel raise test.

mental health (PHQ-9 depression scale, GAD-7 anxiety scale, WHOQOL- BREF quality of life scale, PANAS short form positive and negative affect scale), and perceived global effect of the intervention.

Design:

The study will use a single-group pre-test/post-test design. Participants will be assessed at baseline, after two months of intervention, and at six months follow-up.

Data Analysis:

Data will be analyzed using descriptive statistics and mixed-effects linear regression models.

Significance:

This pilot study will provide valuable information on the feasibility and effect of this group NW intervention for older adults evacuated from their homes. The findings will be used to plan and design a larger longitudinal RCT.

DETAILED DESCRIPTION:
Introduction The outbreak of the Israeli-Hamas conflict on October 7, 2023, triggered widespread displacement, with over 115,000 Israelis evacuated, including 8685 individuals seeking refuge in Haifa. Among these evacuees, older adults face heightened health risks exacerbated, such as PTSD, depression and anxiety, by the trauma of displacement. Evacuation under the threat of war disturb normal living and leads towards a multitude of difficulties spanning various aspects of the evacuees' lives, including economic, environmental, physical and emotional well-being. Studies reveal that maintaining physical activity is crucial for reduction risk of cardiovascular mortality, cancer, recurrent falls, functional and mental decline and maintenance of well-being, yet it becomes challenging amidst the chaos of conflict and relocation.

The WHO recommends 150 minutes of weekly physical activity as a minimum to prevent common health disorders. However, older evacuees, having been displaced from their homes, may struggle to maintain an active lifestyle. After spending four months away from their natural environment, there is a pressing need to reintegrate them into physical activity routines to mitigate potential health risks. Due to the unclear future location of this population, it is important to provide them with the skills, and group support to empower them for sustainable independent walking for the long term.

Nordic walking (NW) is fitness walking with specifically designed poles and a learned technique to create a low stress, total body workout. NW has positive effects on mobility, rehabilitation, and general functioning. In older adults, NW was found effective in improving various age-related disorders: cardiovascular; metabolic; early Parkinson; obesity, and osteoarthritis. NW has also been shown to improve depression, mood, and quality of life.

NW has several biomechanical advantages over walking without poles: it increases gait speed, cardiovascular metabolism, and reduces lower limb and back loads. Increased exercise intensity and energy expenditure that are required in NW are advantageous for older adults to enhance muscle activation and strength. The poles' forward ambulation in NW induces longer steps, and a forceful foot takeoff facilitating higher intensity compared to walking without poles. This study aims to utilize NW benefits for regaining physical activity in a special population at these times of war- the older evacuees.

The proposed Nordic walking group training in Haifa seems to be the first to conduct such a program in Israeli evacuees, and if successful it could be implemented across the country.

The objective of this pilot study is to examine the feasibility of a Nordic walking group intervention to promote sustainable walking, and advance physical and mental health measures in older adults evacuated from their homes to Haifa.

Methods Design: A single-arm, pre-post-intervention. Ethics was approved by the Faculty's Ethics committee (Application no. ECH043693). The investigators plan to launch the first group on May 2024. Population: An exposure meeting was conducted on March 17th for the older adults from Kibutz Dan, and 31 registered to participate, age of 65+ years, free walking ability, medical approval by GP to participate.

The intervention will consist of 60-minute NW group sessions, twice weekly, for two months (total 16 sessions). Participants will be provided with NW sticks to use during the sessions. Each NW session will be led by a qualified healthcare professional that received 4 hours NW guidance qualification, and participated in 4 sessions prior to leading one. Current qualified healthcare professionals are 2 physiotherapists (HSB, HI), and a nurse (LKG). Final year physiotherapy students will assist the lead trainer, hence each session will be guided by two members of the research team- a clinician and a graduating student.

A social worker (SP) will participate in one weekly session aiming to empower the participants and utilize group dynamics techniques to promote successful continuation of independent walking following the guided period. SP will observe the members during training, and converse with them informally (no structured interviews will be included) to identify suitability for roles within the group, such as leading, supporting, adhering etc.

Communication throughout the study will be conducted via a WhatsApp forum, to motivate and sustain regular walking during and after the training period. Following 2 months of guidance the group will be launched independently, while keeping remote contact. Same frequency and schedule will be encouraged.

Procedure: All recruited participants will provide informed consent prior to their enrollment. Assessments will be conducted at baseline, following 2 months of guided sessions, and follow up after additional 2 and 4 months (total 6 months procedure).

Primary measures: (1) Adherence with independent walking for at least 150 minutes per week, over 4 months follow up. Optimal adherence outcome will be up to 20% absence. (2) Steps count- via a mobile application, will provide an objective quantified measure of walking. Secondary measures are detailed in the relevant section.

Data analysis The Friedman test will be used to compare Adherence across the time points (pre-, post-intervention, follow-up). A post hoc Wilcoxon signed-rank test will be conducted if the overall test shows significance with a Bonferroni correction to multiple testing. Significance levels will be set at 0.05. JMP and SPSS software will be used for statistical analysis.

In summary, this is one of the most challenging periods in Israeli history. For over four months, thousands of older Israelis have been evacuated from their homes. Providing Nordic walking to this population is an evidence based, effective, and safe training to provide them with. They need our assistance to prevent deuteriation of their mental and physical health.

After establishing the most effective format to sustain independent safe walking in older evacuees, the investigators will be able to expand it to the rest of the country - walking together for a better tomorrow.

Time plan: Planning, set up, trainers' qualification, and ethics revisions are in final stages at present. Data collection- 6 months; Data analysis- 3 months; Write up of findings for publication in Q1-2 journal- 3 months; Total duration- 12 months

Scope of Impact Our pilot study will help us determine whether the timeline to independence can be achieved, how to empower the group, barriers to compliance and adherence, and how to collect outcome measures efficiently. The investigators will be able to extend the customized model of this NW program to all hotels in Haifa, and if successful- to the rest of the country. Any older adult community could benefit from this model, so it may be applicable globally.

This is a collaborative study proposal between the Department of Physiotherapy and Gerontology in the University of Haifa and the Haifa district health bureau. This model, if found effective and beneficial, can be exported to other districts in Israel in collaboration with the Ministry of Health.

ELIGIBILITY:
Inclusion Criteria:

* Participants in stable health and have been cleared by their doctor to participate in physical activity.

Exclusion Criteria:

* Using an assisting device for walking
* Any health condition that may prevent participants from doing physical activity according to their medical doctor.
* Unstable gait with high risk of fall by subjective and physical assessment,
* Dizziness, visual or hearing impairment that cannot be corrected.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Steps count by a smartphone application. | Baseline; immediately after intervention completion (week 8); 2,4 months post intervention follow-up.
  weakly and monthly average of steps count will be retrieved from the cellular application.
Adherence (number of patients that attended training sessions during the intervention time and throughout 4 months post intervention) | participation will be monitored during the 8 weeks of intervention. Follow up evaluation of independent walking throughout 4 months after intervention completion.
  Adherence to the walking program: participation in the 16 trained sessions during the intervention, and adherence to 150min/week during follow up period of 4 months post intervention. Optimal adherence outcome will be up to 20% absence.

SECONDARY OUTCOMES:
30 seconds Sit to stand test (number of repetitions for measuring lower limb strength and balance) | Baseline; immediately after intervention completion (week 8); 2,4 months post intervention follow-up.
  30 Seconds Sit to Stand Test is a validated functional measure for lower limb strength and balance. Evidence-based threshold values indicate risk of fall are dependent on age and gender function (30-second sit-to-stand test, heel raise test, 4-meter walk test), mental health (PHQ-9 depression scale, GAD-7 anxiety scale, WHOQOL- BREF quality of life scale, PANAS short form positive and negative affect scale), and perceived effectiveness of the intervention.
Two-minute walk test ( distance in meters for measuring functional endurance and gait performance) | Baseline; immediately after intervention completion (week 8); 2,4 months post intervention follow-up.
  The two-meter Walk Test is a validated test for measuring functional endurance and assessing gait performance in older adults.
Patient Health Questionnaire (score in depression questionnaire to assess the risk of developing mental health problems) | Baseline; immediately after intervention completion (week 8); 2,4 months post intervention follow-up.
  A nine-item depression questionnaire. PHQ-9 would help to identify individuals who may be at risk of developing mental health problems. The scale ranges from 0-27, a high score means worse outcome.
Generalized Anxiety Disorder (score in anxiety questionnaire to assess the risk of developing mental health problems) | Baseline; immediately after intervention completion (week 8); 2,4 months post intervention follow-up.
  A seven-item generalized anxiety disorder questionnaire. GAD-7 would help to identify individuals who may be at risk of developing mental health problems. The scale ranges from 0-21, a high score means worse outcome.
The World Health Organization quality of life assessment (score in the questionnaire to assess quality of life) | Baseline; immediately after intervention completion (week 8); 2,4 months post intervention follow-up.
  The World Health Organization quality of life assessment (WHOQOL-Bref) is the most frequently used measure to evaluate Quality of life in displaced populations. The scale ranges from 2-10, a high score means a better outcome.
The Positive and Negative Affect Schedule (score in the questionnaire to assess mood) | Baseline; immediately after intervention completion (week 8); 2,4 months post intervention follow-up.
  The Positive and Negative Affect Schedule (PANAS) is a 10-item scale for measuring positive and negative affect. The scale ranges from 5-25 for both positive and negative feelings, separately. A better outcome means a high score in positive affect and a low score in negative affect. It was found reliable, valid, and efficient means for measuring these two important dimensions of mood.
Global perceived effect (score in the questionnaire to assess perceived effect of the NW intervention) | immediately after intervention completion (week 8); 2,4 months post intervention follow-up.
  Global perceived effect (GPE), is an 11-point scale to assess the perceived effect of the NW intervention (-5 worst negative effect, 0=no effect, +5 best positive effect).
Heel Raise Test (number of repetitions for measuring ankle plantarflexion strength) | Baseline; immediately after intervention completion (week 8); 2,4 months post intervention follow-up.
  The ankle plantar flexor muscles are contributors to the performance of many mobility activities including sit-to-stand, walking, running and climbing stairs. As a result, Quantifying the muscles' strength is important.

CONTACTS AND LOCATIONS:
Overall Officials: Hilla Sarig-Bahat, Phd, Principal Investigator — University of Haifa, Haifa, Israel
Locations (1):
- Dan Carmel Hotel, Haifa, Israel

REFERENCES:
- [Background] Cantor D, Swartz J, Roberts B, Abbara A, Ager A, Bhutta ZA, Blanchet K, Madoro Bunte D, Chukwuorji JC, Daoud N, Ekezie W, Jimenez-Damary C, Jobanputra K, Makhashvili N, Rayes D, Restrepo-Espinosa MH, Rodriguez-Morales AJ, Salami B, Smith J. Understanding the health needs of internally displaced persons: A scoping review. J Migr Health. 2021 Oct 29;4:100071. doi: 10.1016/j.jmh.2021.100071. eCollection 2021. PMID 34820657
- [Background] Ding D, Mutrie N, Bauman A, Pratt M, Hallal PRC, Powell KE. Physical activity guidelines 2020: comprehensive and inclusive recommendations to activate populations. Lancet. 2020 Dec 5;396(10265):1780-1782. doi: 10.1016/S0140-6736(20)32229-7. Epub 2020 Nov 25. No abstract available. PMID 33248019
- [Background] The World Health Organization Quality of Life assessment (WHOQOL): position paper from the World Health Organization. Soc Sci Med. 1995 Nov;41(10):1403-9. doi: 10.1016/0277-9536(95)00112-k. PMID 8560308
- [Background] Phraknoi N, Sutanto J, Hu Y, Goh YS, Lee CEC. Older people's needs in urban disaster response: A systematic literature review. International Journal of Disaster Risk Reduction. 2023:103809.
- [Background] Ben Simon B, Toporek Barr O, Kermel-Schiffman I, Sorek Y, Resnizky S, Jacobovitz Y. The Israel-Hamas War - The Impact of Loss and Bereavement on Families and the Community: A Litererature Review. In: Shani M, ed. Jerusalem, Israel: Myers JDC Brookdale Institute; 2023.
- [Background] Swanson CW, Haigh ZJ, Fling BW. Two-minute walk tests demonstrate similar age-related gait differences as a six-minute walk test. Gait Posture. 2019 Mar;69:36-39. doi: 10.1016/j.gaitpost.2019.01.019. Epub 2019 Jan 14. PMID 30660949
- [Background] Bohannon RW, Wang YC, Gershon RC. Two-minute walk test performance by adults 18 to 85 years: normative values, reliability, and responsiveness. Arch Phys Med Rehabil. 2015 Mar;96(3):472-7. doi: 10.1016/j.apmr.2014.10.006. Epub 2014 Oct 25. PMID 25450135
- [Result] Cunningham C, O' Sullivan R, Caserotti P, Tully MA. Consequences of physical inactivity in older adults: A systematic review of reviews and meta-analyses. Scand J Med Sci Sports. 2020 May;30(5):816-827. doi: 10.1111/sms.13616. Epub 2020 Feb 4. PMID 32020713
- [Result] Wang Z, Jiang B, Wang X, Li Z, Wang D, Xue H, Wang D. Relationship between physical activity and individual mental health after traumatic events: a systematic review. Eur J Psychotraumatol. 2023;14(2):2205667. doi: 10.1080/20008066.2023.2205667. PMID 37134018
- [Result] Russo L, Belli G, Di Blasio A, Lupu E, Larion A, Fischetti F, Montagnani E, Di Biase Arrivabene P, De Angelis M. The Impact of Nordic Walking Pole Length on Gait Kinematic Parameters. J Funct Morphol Kinesiol. 2023 Apr 26;8(2):50. doi: 10.3390/jfmk8020050. PMID 37218846
- [Result] Skorkowska-Telichowska K, Kropielnicka K, Bulinska K, Pilch U, Wozniewski M, Szuba A, Jasinski R. Nordic walking in the second half of life. Aging Clin Exp Res. 2016 Dec;28(6):1035-1046. doi: 10.1007/s40520-016-0531-8. Epub 2016 Jan 23. PMID 26803510
- [Result] Bieler T, Siersma V, Magnusson SP, Kjaer M, Christensen HE, Beyer N. In hip osteoarthritis, Nordic Walking is superior to strength training and home-based exercise for improving function. Scand J Med Sci Sports. 2017 Aug;27(8):873-886. doi: 10.1111/sms.12694. Epub 2016 Apr 30. PMID 27129607
- [Result] Liu Y, Xie W, Li J, Ossowski Z. Effects of aerobic exercise on metabolic indicators and physical performance in adult NAFLD patients: A systematic review and network meta-analysis. Medicine (Baltimore). 2023 Apr 7;102(14):e33147. doi: 10.1097/MD.0000000000033147. PMID 37026928
- [Result] Gobbo S, Bullo V, Roma E, Duregon F, Bocalini DS, Rica RL, Di Blasio A, Cugusi L, Vendramin B, Bergamo M, Cruz-Diaz D, Alberton CL, Ermolao A, Bergamin M. Nordic Walking Promoted Weight Loss in Overweight and Obese People: A Systematic Review for Future Exercise Prescription. J Funct Morphol Kinesiol. 2019 Jun 18;4(2):36. doi: 10.3390/jfmk4020036. PMID 33467351
- [Result] Rodrigues IB, Ponzano M, Butt DA, Bartley J, Bardai Z, Ashe MC, Chilibeck PD, Thabane L, Wark JD, Stapleton J, Giangregorio LM. The Effects of Walking or Nordic Walking in Adults 50 Years and Older at Elevated Risk of Fractures: A Systematic Review and Meta-Analysis. J Aging Phys Act. 2021 Oct 1;29(5):886-899. doi: 10.1123/japa.2020-0262. Epub 2021 Feb 11. PMID 33571958
- [Result] Kyrdalen IL, Thingstad P, Sandvik L, Ormstad H. Associations between gait speed and well-known fall risk factors among community-dwelling older adults. Physiother Res Int. 2019 Jan;24(1):e1743. doi: 10.1002/pri.1743. Epub 2018 Sep 10. PMID 30198603
- [Result] Roongbenjawan N, Siriphorn A. Accuracy of modified 30-s chair-stand test for predicting falls in older adults. Ann Phys Rehabil Med. 2020 Jul;63(4):309-315. doi: 10.1016/j.rehab.2019.08.003. Epub 2019 Sep 11. PMID 31520784
- [Result] Bohannon RW. The heel-raise test for ankle plantarflexor strength: a scoping review and meta-analysis of studies providing norms. J Phys Ther Sci. 2022 Jul;34(7):528-531. doi: 10.1589/jpts.34.528. Epub 2022 Jul 1. PMID 35784604
- [Result] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Result] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Result] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Result] Gagliardi J, Brettschneider C, Konig HH. Health-related quality of life of refugees: a systematic review of studies using the WHOQOL-Bref instrument in general and clinical refugee populations in the community setting. Confl Health. 2021 Jun 2;15(1):44. doi: 10.1186/s13031-021-00378-1. PMID 34078413
- [Result] Kamper SJ, Ostelo RW, Knol DL, Maher CG, de Vet HC, Hancock MJ. Global Perceived Effect scales provided reliable assessments of health transition in people with musculoskeletal disorders, but ratings are strongly influenced by current status. J Clin Epidemiol. 2010 Jul;63(7):760-766.e1. doi: 10.1016/j.jclinepi.2009.09.009. Epub 2010 Jan 8. PMID 20056385
- [Result] Liu Y, Xie W, Ossowski Z. The effects of Nordic Walking on health in adults: A systematic review. Journal of Education, Health and Sport. 2023;13:188-196.